CLINICAL TRIAL: NCT04949321
Title: Acceleration of the Kinetics of Diffusion of Gadolinium in the Perilymphatic Structures of the Inner Ear.
Acronym: FAST-HYDROPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 38RC20.394
Record Dates: First submitted 2021-06-24; First posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Inner Ear ; Meniere's Disease; Imaging
Keywords: Magnetic Resonance Imaging; Contrast Media
MeSH Terms: conditions — Meniere Disease | interventions — Magnetic Resonance Spectroscopy; gadobutrol

STUDY DESIGN:
Masking Description: 60 Meniere's Disease patients and 20 healthy volunteers (sample of 5 volunteers per MRI machine)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gadovist (gadobutrol) / two MRI (Experimental): 60 Meniere's Disease patients and 20 healthy volunteers (sample of 5 volunteers per MRI machine)
  Interventions: Other: Magnetic Resonance Imaging with Single dose of gadobutrol (Gd-DO3A-butrol, Gadovist® 0.1 mmol/kg, 1 mmol/mL)

INTERVENTIONS:
Other: Magnetic Resonance Imaging with Single dose of gadobutrol (Gd-DO3A-butrol, Gadovist® 0.1 mmol/kg, 1 mmol/mL) — Magnetic Resonance Imaging with Single dose of gadobutrol (Gd-DO3A-butrol, Gadovist® 0.1 mmol/kg, 1 mmol/mL)

SUMMARY:
To determine the optimal delay after Gadolinium injection to analysis inner ear structures as measured by repeated MR 3D-FLAIR Weighted Imaging. We hypothesize that the endolymphatic structures can be distinguished earlier than 4 hours after contrast media injection.

DETAILED DESCRIPTION:
The gadolinium contrast agents are now required to cross the blood-perilymph inner ear barrier after an intravenous administration in order to assess the endolymphatic structures in patients with vertigo or hearing loss, using MRI with delayed acquisition (at least 4 hours between injection and images acquisition).

This technique relies on the glymphatic diffusion of the gadolinium agents (Naganawa et al.,MRM Sci 2017) and has proved to be useful in patients with Meniere's Disease (Naganawa et al., AJNR 2014, Attyé et al., Eur Radiol 2018), Recurrent Peripheral Vestibulopathy (Attye et al., Eur Radiol 2015) or Otosclerosis (Mukaida et al., Otol Neurotol 2015), leading to numerous scientific publications over the last decade. The inner ear perilymph enhancement is particularly important to distinguish the saccule from the utricle, these inner ear structures were recently used to classify with imaging Meniere's Disease patient (Attye et al; European Radiology 2016).

We recently demonstrated in patients (Eliezer et al., J Neuroradiol 2018), comparing the effect of two macrocyclic contrast agents (Gd-DOTA, Dotarem® and Gd-DO3A-butrol, Gadovist®), that the Gd-DO3A-butrol better enhanced inner ear structures that Gd-DOTA, both with qualitative and quantitative analysis, allowing to more accurately diagnose endolymphatic hydrops in Meniere's Disease patients.

We have speculated that the differences in the physiochemical properties of Gd-contrast agents (concentration, relaxivity, osmalality) are determining factors to cross the blood-perilymph barrier.

These properties should allow scanning diseased patients earlier after contrast media administration, the delay between the injection and MRI acquisition being actually a limitation to expand this technique in the clinical setting, particularly with 1.5T magnets, due to the low Signal to Noise Ratio using 3D-FLAIR sequences analysis.

Here, we want to conduct multi-centre prospective clinical and radiological study to determine the optimal timing to explore Meniere's Disease patient after Gadobutrol injection with single dose intravenous administration.

ELIGIBILITY:
Inclusion criteria; Healthy volunteers Major subjects of over 40 years (mean age of Meniere's disease 40 to 50 years) Informed consent signed Medical examination performed prior to participation in research Patients without history of inner ear disease

Meniere's Disease Major subjects of over 40 years (mean age of Meniere's disease 40 to 50 years) Informed consent signed Medical examination performed prior to participation in research Patients with clinical criteria of Meniere's disease according to the classification of the American Association of Otology (ie the combination of a sensorineural hearing loss at low frequencies, recurrent vertigo and tinnitus and / or clogged ear sensation)

Exclusion criteria:

Patients minors Patients pregnant Patients on a legal protection regime type guardianship Respiratory pathologies, cardiovascular or renal disorders, neurological diseases Claustrophobia Contraindications to exposure to a magnetic field Contraindications to injecting Gadovist® Other ongoing clinical trials with exclusion period for MRI

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-07-31 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Adapted visualization of the saccule and utricle on the early MR sequences when compared to the 4-hours MR 3D FLAIR sequence (gold standard). | 4 hours
  Qualitative:Visibility/Visual evaulation of the endolymphatic structures (saccule/utricle) on various 3D-FLAIR acquisition
  For endolymphatic hydrops analysis, we will use the classification that we have published in European Radiology (Attye et al, Eur Radiol 2016).
  Quantitative: T1 mapping: Automatic and manual measurement of the T1 relaxation time values of the endolymph for each MR sequence by drawing ROIs.

SECONDARY OUTCOMES:
Gadolinium enhancement in basal nuclei as measured by T1 and T2 relaxometry maps. | 4 hours
  T1 mapping: Automatic and manual measurement of the T1 relaxation time values of the endolymph for each MR sequence by drawing ROIs.